CLINICAL TRIAL: NCT04277923
Title: Effects of Medium and Long Chain Fat Emulsions and SMOF Fat Emulsions on PNALD and Oxidative Stress in Premature Infants: a Randomized, Double-blind Controlled Study
Brief Title: Effects of Fat Emulsions on PNALD and Oxidative Stress in Premature Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ying Wang, head of department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PNALD
Record Dates: First submitted 2020-01-06; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Preterm Infant
Keywords: parenteral nutrition; lipid emulsion; SMOF; PNALD; oxidative stress
MeSH Terms: conditions — Premature Birth; Hyperphagia | interventions — SMOFlipid; Lipofundin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMOF lipid emulsion (Experimental): the SMOF lipid emulsion is SMOFlipid.
  Interventions: Drug: SMOFlipid
- MCT/LCT lipid emulsion (Experimental): the MCT/LCT lipid emulsion is Lipofundin.
  Interventions: Drug: Lipofundin

INTERVENTIONS:
Drug: SMOFlipid — the lipid of all-in-one is less than 4g/kg.d
  Arms: SMOF lipid emulsion
Drug: Lipofundin — the lipid of all-in-one is less than 4g/kg.d
  Arms: MCT/LCT lipid emulsion

SUMMARY:
Abnormal liver function or cholestasis is the result of multiple factors, include low birth weight, smaller than gestational age, preterm birth, infection, lipid emulsion (LE) in parenteral nutrition (PN), insufficient enteral nutrition (EN) etc. Most are inevitable, but the LEs in PN can be selected. So the investigators compare two LEs, and want to see if the SMOF LE can improve hepatic index in preterm infants.

DETAILED DESCRIPTION:
For preterm infants, especially for very or extremely low birth weight infants, it's impossible to achieve total enteral feeding in short time. So, PN has played an important role to sustain normal life. But, it also has an adverse effect on liver namely parenteral nutrition-associated liver disease (PNALD). LE(s) in PN has been showed to result in PNALD. So changing the type of LEs has been an ideal solution.

Two types of lipid emulsions are currently used for pediatric patients: one LE(the second generation) is composed of 50% long-chain triacylglycerols (LCTs) and 50% medium-chain triacylglycerols (MCTs), prepared from soybean oil and coconut oil respectively. A new LE (SMOF) contains 30% LCTs, 30% MCTs, 25% olive oil, and 15% fish oil. SMOF is rich in omega-3 polyunsaturated fatty acids which derived from fish oil. It may reduce inflammation in premature infants, prevent or treat cholestasis, and reduce oxidative stress.

Because of the different compositions, they have different effect on liver, inflammation, oxidative stress, etc. Therefore, the investigators designed a prospective, randomized and double-blind study to compare the different LEs (MCTs/LCTs and SMOF), so as to select a more suitable fat emulsion for premature infants in order to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (gestational age < 32 weeks) with birth weight < 1500g were admitted to NICU of Xin Hua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China within 24 hours after birth
* No contraindications to parenteral nutrition
* Expected PN support for 14 days or more
* Parents or guardians agree

Exclusion Criteria:

* Parenteral nutrition support was provided prior to enrollment
* EN calorie for 10% or more
* Congenital intestinal structural/functional abnormalities
* Liver function damage caused by viral hepatitis, genetic metabolism and abnormal biliary tract
* Congenital or acquired immunodeficiency
* Complex congenital heart disease

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change of liver function indexes | change from baseline in liver function indexes at 7 days and 14 days
  liver enzyme in u/L
Change of bilirubin indexes | change from baseline in bilirubin indexes at 7 days and 14 days
  bilirubin in μmol/L

SECONDARY OUTCOMES:
Change of superoxidase dismutase | change from baseline in superoxidase dismutase at 7 days and 14 days
  superoxidase dismutase in u/L
Change of malondialdehyde | change from baseline in malondialdehyde at 7 days and 14 days
  malondialdehyde in nmol/ml
Change of inflammatory factors | change from baseline in fatty acid at 7 days and 14 days
  IL-1B, IL-2R, IL-6, IL-8, IL-10 and TNF-α in pg/ml

OTHER OUTCOMES:
Change of fatty acids spectrum | change from baseline in fatty acids spectrum at 7 days and 14 days
  cholic acid, deoxycholic acid,chenodeoxycholic acid,ursodeoxycholic acid and lithocholic acid in mol%,et al.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Phd, Principal Investigator — Xin Hua Hospital, School of Medicine, Shanghai Jiao Tong University,China